CLINICAL TRIAL: NCT01331057
Title: Validation of "AVICENNE's ELAL": Instrument of Mother Tongue Assessment and Impact of Familial and Transcultural Factors on Early Bilingualism in Migrants' Children Born in France
Brief Title: Bilingualism: Validation Of "Avicenne's Elal"
Acronym: BILINGUISME
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: NI07023
Record Dates: First submitted 2011-04-05; First posted 2011-04-07 (Estimated); Last update posted 2021-06-15 (Actual); Status verified 2021-06

CONDITIONS: Language
Keywords: Bilingualism; Language; Evaluation transcultural; Intra Familial Relationship; Transmissions mother; Tongue french; Language tamil; Language arabic; Language soninke; Language cultural; Affiliations crossbreeding
MeSH Terms: conditions — Language | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1:Sri Lankais: Children aged of four to six years old, in the nursery school and if their first language is unique : tamil.
  Interventions: Other: NEEL test; Other: ELAL test; Other: Interview
- 2: Algerian: Children aged of four to six years old, in the nursery school and if their first language is unique : arabic.
  Interventions: Other: NEEL test; Other: ELAL test; Other: Interview
- 3: Mali: Children aged of four to six years old, in the nursery school and if their first language is unique : SONINKE.
  Interventions: Other: NEEL test; Other: ELAL test; Other: Interview

INTERVENTIONS:
Other: NEEL test — An assessment for children in French with items extracted from the NEEL test
Other: ELAL test — An assessment of mother tongue with the ELAL of AVICENNE
Other: Interview — For parents of children include in the study: A semi -structured interview

SUMMARY:
The primary purpose is the validation of an instrument of the first language assessment. The second purpose is to study the impact of familial and transcultural factors on early bilingualism in migrant children born in France.

DETAILED DESCRIPTION:
The research aims to validate a language instrument of the first language in migrants' children born in France. For that purpose, the investigators have built an instrument made of three sets of items: comprehension, production and narrative production. Children are elected if: they are four to six years old, in the third class of nursery school and if their first language is unique, and, one of the three languages that the investigators define for the first step of validation: tamil, SONINKE, Arabic. The PROTOCOLE is composed with two parts:

1. For children:

   * An assessment for children in French with items extracted from the NEEL test
   * An assessment of mother tongue with the ELAL of Avicenne
2. For parents:

   * A semi-structured interview.

The data collected are:

General DATA:

* Social and professional categories
* Economical status of parents
* The conditions of living
* Month and year of birth for the child
* The language used during the interview

About the child:

* Age of language AQUISITION
* Languages mastering
* Language environment
* The place among siblings
* SCOLARISATION(DATA about cultural affiliations, representations of transmission, intra-familial relationship

DATA about parental uses and representations of languages:

* Social and economical DATA in the country of birth
* Place of birth, languages
* uses of languages
* representations about languages

ELIGIBILITY:
Inclusion Criteria:

* Age : four to six years old
* SCOLARISATION : nursery school
* One language in the family house: tamil, Arabic, or SONINKE

Exclusion Criteria:

* first class of elementary school
* two mother tongues in the family

Ages: 5 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children are five to six years old, in the third class of nursery school and if their first language is unique, and, one of the three languages that we defines for the first step of validation: tamil, soninké, Arabic
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2011-06 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Validation of an instrument of the first language assessment. | at 54 months
  Validation of "avicenne's ELAL": instrument of mother tongue assessment

SECONDARY OUTCOMES:
Impact of familial and transcultural factors | at 54 months
  impact of familial and transcultural factors on early bilingualism in migrants' children born in france

CONTACTS AND LOCATIONS:
Overall Officials: Dalila REZZOUG, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Dr Dalila REZZOUG, Bobigny, Seine Saint-Denis, France